CLINICAL TRIAL: NCT05754203
Title: Efficacy and Safety of Super-hyperfractionation Pulse Radiotherapy Combined With Immune Checkpoint Inhibitor for Advanced Non-small Cell Lung Cancer.
Brief Title: Efficacy and Safety of Super-hyperfractionation Pulse Radiotherapy Combined With ICIs for Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director of oncology department, Clinical Professor, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-020
Record Dates: First submitted 2023-02-12; First posted 2023-03-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Immune Checkpoint Inhibitor; Radiotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Super-hyperfractionation Pulse Radiotherapy Combined With Immune Checkpoint Inhibitor (Experimental): Radiotherapy design: a single dose of 0.5Gy, 16 consecutive pulses with an interval of 3 minutes (0.5Gy * 16F), total dose DT: 8Gy; Immunotherapy: PD-1/PD-L1 monoclonal antibodies conforming to CSCO guidelines for lung cancer indications, including Carrilizumab, Tirelizumab, Teripril, Paborizumab, etc., conventional therapeutic dose, Q3W, until progression or the investigator judges that there is no longer clinical benefit or intolerable side effects.
  Interventions: Radiation: Super-hyperfractionation Pulse Radiotherapy

INTERVENTIONS:
Radiation: Super-hyperfractionation Pulse Radiotherapy — Radiotherapy design: a single dose of 0.5Gy, 16 consecutive pulses with an interval of 3 minutes (0.5Gy * 16F), total dose DT: 8Gy; Immunotherapy: PD-1/PD-L1 monoclonal antibodies conforming to CSCO guidelines for lung cancer indications, including Carrilizumab, Tirelizumab, Teripril, Paborizumab, etc., conventional therapeutic dose, Q3W, until progression or the investigator judges that there is no longer clinical benefit or intolerable side effects.
  Other Names: Immune Checkpoint Inhibitor

SUMMARY:
Investigators intend to combine low-dose hypersensitivity with high-dose immunopotentiation effect, and use super-hyperfractionation pulse radiotherapy, which is expected to achieve the effect of in situ vaccine that can enhance tumor killing, protect normal tissues, reduce immune cell damage and enhance tumor immunogenicity at the same time, and play a stronger immunopotentiation effect in combined immunotherapy. Thereby inducing a stronger abscopal effect of radiotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Informed consent has been signed and, in the judgment of the investigator, the patient is able to comply with the study protocol and sign a written informed consent.
2. Participants diagnosed with stage IIIB or above non-small cell lung cancer confirmed by histopathology (whether newly diagnosed or not) meet the requirements of SBRT radiotherapy (mass limited, less than 5 cm) and immune checkpoint inhibitor therapy (according to CSCO guidelines).
3. Age ≥ 18 and less than 75.
4. Eastern Cooperative Oncology Group Performance Status Score (ECOG PS) 0-3.

Exclusion Criteria

1. The participant's compliance is poor and the test regulations are violated.
2. Dysfunction of important organs of liver and kidney, such as myocardial infarction, angina pectoris, and significant increase of liver transaminase.
3. Any disease requiring systemic treatment with corticosteroids or other immunosuppressive drugs within 14 days prior to enrollment.
4. Serious infection within 4 weeks before enrollment, including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia.
5. Severe chronic or active infections (including tuberculosis infection) requiring systemic (oral or intravenous) antibiotic therapy within 14 days before enrollment.
6. Participants with untreated chronic hepatitis B or HBV carriers with hepatitis B virus (HBV) DNA ≥ 500 IU/mL, or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B, HBsAg carriers, treated and stable hepatitis B carriers (HBV DNA < 500 IU/mL), and cured hepatitis C patients can be included in the group.
7. Known history of HIV infection.
8. Receive any other investigational drug treatment or participate in other clinical trials within 28 days.
9. There are no contraindications to stereotactic radiotherapy and immune checkpoint inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 12 weeks
  The proportion of patients with tumor volume reduced by 30% and maintained for more than 4 weeks. Sum of the proportions of complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
iORR | 24 weeks
  The objective response rate away from the radiation field

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Sun, Principal Investigator — Department of Oncology, Xinqiao Hospital, Army Medical University
Locations (2):
- China (2):
  - the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality
  - Jianguo Sun, Chongqing

IPD SHARING:
Plan to Share IPD: No